CLINICAL TRIAL: NCT00001953
Title: Basal and Stimulated Somatostatin Plasma Levels in Patients With Primary Sjogren's Syndrome and in Control Subjects
Brief Title: The Functioning of Immune and Hormonal Systems in Patients With Sjogren's Syndrome and in Healthy Volunteers
Status: Completed | Type: Observational
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000022; 00-D-0022
Record Dates: First submitted 2000-01-18; First posted 2000-01-19 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2001-12

CONDITIONS: Sjogren's Syndrome
Keywords: Endocrine System; Autoimmunity; Salivary Glands; Glucose Tolerance Test; Growth Hormone; Somatostatin; Sjogren's Syndrome
MeSH Terms: conditions — Sjogren's Syndrome; Autoimmune Diseases

SUMMARY:
This study aims to learn more about how the immune and hormonal systems function in patients with Sjogren's syndrome, a disease in which the immune system does not function properly. Adult nonpregnant females are invited to participate. Oral contraceptives may not be taken for 6 weeks before and during this study, so another form of birth control must be used, such as abstinence.

There will be two visits. At the first visit, a medical history and physical examination will be conducted, and blood and urine tests will be done. The total amount of blood drawn will be 10 tablespoons. This visit will last 3 hours. At the second visit, participants will have an oral glucose tolerance test. To prepare for it, they must be on a special diet for 3 days beforehand and keep a diary of eating, sleeping, and physical activities for those 3 days. A urine sample will be taken at the beginning of the visit. Subjects must then drink a very sweet carbonated cola. A small plastic tube will be placed into an arm vein. Blood will be drawn through this tube eight times over 3 hours. The total amount of blood drawn will be 17 tablespoons.

Only minor inconveniences are anticipated as a result of participating in this study. Risks from blood tests include soreness, bruising, and minor infection at the puncture site, and dizziness. The oral glucose tolerance test may cause temporary stomach bloating, headache, nausea, and vomiting.

DETAILED DESCRIPTION:
Sjogren's syndrome is a chronic systemic disease that primarily affects the salivary and lacrimal glands and is characterized by lymphocytic tissue infiltration and auto-antibody production. The pathogenesis of Sjogren's syndrome is unknown. We hypothesize that reduced somatostatin activity is an important factor in promoting immune dysregulation in patients affected by Sjogren's syndrome. Somatostatin is a multifunctional peptide with potent immunomodulatory properties whose effects are reduced lymphocytic activity, reduced gastrointestinal secretions, activation of the hypothalamic-pituitary axis, anti-inflammatory, etc. As several findings in Sjogren's syndrome are opposite to those produced by somatostatin, it is logical to consider that the activity of this peptide is low in patients affected by this disease. The purpose of this study is to determine whether basal and stimulated plasma levels of somatostatin and its effects on the immune and endocrine systems differ between 16 patients affected by primary Sjogren's syndrome and 16 healthy control subjects.

ELIGIBILITY:
Female gender only, ages 18 to 75.

Patients should have documented primary Sjogren's syndrome as determined by protocol 84-D-0056. The diagnosis of primary Sjogren's syndrome will be based on the presence of all three of the following:

Salivary gland abnormalities;

Lacrimal gland abnormalities;

Serologic abnormalities.

Controls should have no signs or symptoms of Sjogren's syndrome, and negative serologic testing reconfirmed within 2 weeks of the OGTT.

Willingness to: a) participate in phase I and II of the protocol; b) follow the guidelines set to prepare for the OGTT; and c) modify current medical therapy if necessary.

Must be able to comply with protocol procedures.

No patients with "incomplete" Sjogren's syndrome, i.e., with less than three positive findings as described above.

No presence of physical or mental conditions that may interfere with the protocol. These include the following diseases and conditions:

(Present at time of phase I/II): significant disruption of sleep-wake pattern (i.e., less than 4 hours of continuous sleep, on the night before the OGTT only), BMI less than 18 or equal to/greater than 30, anemia with Hgb less than 10 gm/dl, use of tobacco or alcohol;

(Within the past 6 weeks): acute weight change (greater than 5%), use of contraceptives -BCP-, Depoprovera or Norplant), irregular menstrual cycle, lactation, blood drawing in excess of 50 ml, use of recreational drugs, modification of estrogen replacement therapy;

(Within the past 6 months): chronic pattern of weight change (greater than 10%), eating disorders, uncontrolled hypo/hyperthyroidism, breast cancer, lymphoma or other malignancy, pregnancy, treatment for depression, insulinoma, VIPoma, pheochromocytoma, atrophic gastritis, active tuberculosis or treatment for it;

(A history of): HIV+, sarcoidosis, secondary Sjogren's syndrome, bleeding diathesis, organ transplant, severe neuroendocrine, renal, cardiovascular, pulmonary or gastrointestinal disease (e.g., renal insufficiency, unstable angina, heart failure, severe emphysema, Crohn's disease), diabetes mellitus, acromegaly and mental retardation.

No contraindications to OGTT. These include:

Hospital inpatient status, acute illness, immobilization, starvation, severe emotional distress within one week of the OGTT;

Low carbohydrate diet (less than 150 g/day) for 3 days preceding the OGTT;

Pregnancy;

Therapy which impairs glucose tolerance: e.g., niacin, thiazide diuretics, phenytoin, excess thyroxine or psychotropic drugs within 1 month of phase I, oral contraceptives within 6 weeks of phase I, glucocorticoid treatment within the past 6 months (or one year if treatment lasted over 2 weeks), Beta blockers/agonists (e.g., terbutaline) within 2 days of phase I;

Diabetes mellitus;

Glucose intolerance.

Subjects may not take medications that can affect somatostatin levels, such as antidepressants, benzodiazepines, neuromodulators (e.g., cholinergic, alpha/beta adrenergic), oral contraceptives (BCP), steroid hormones (with the exception of estrogen replacement therapy -ERT-, for which subjects will be matched), immunomodulators, anticonvulsants (e.g., carbamazepine), cimetidine -Tagamet® (Registered Trademark)-, herbal remedies (because of their variable substance content). Subjects may not take drugs affecting gastrin secretion: antacids (e.g., Maalox® (Registered Trademark), Mylanta® (Registered Trademark), H(2) receptor antagonists (e.g., famotidine -Pepcid® (Registered Trademark)-, ranitidine -Zantac® (Registered Trademark)-), cathecolamines, atropine, haloperidol. To become eligible, subjects should be able to safely discontinue these medications at least one month prior to phase I. Antacids, H(2) antagonists and neuromodulators (e.g., Salagen) may be discontinued 2 days prior to phase I.

Patients cannot have take experimental drugs within 1 month of the beginning of the protocol.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32
Dates: Start 1999-11; Study Completion 2001-12

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Dental And Craniofacial Research (NIDCR), Bethesda, Maryland, United States

REFERENCES:
- [Background] Fox RI, Tornwall J, Maruyama T, Stern M. Evolving concepts of diagnosis, pathogenesis, and therapy of Sjogren's syndrome. Curr Opin Rheumatol. 1998 Sep;10(5):446-56. doi: 10.1097/00002281-199809000-00009. PMID 9746861
- [Background] Fox PC, Speight PM. Current concepts of autoimmune exocrinopathy: immunologic mechanisms in the salivary pathology of Sjogren's syndrome. Crit Rev Oral Biol Med. 1996;7(2):144-58. doi: 10.1177/10454411960070020301. PMID 8875029
- [Background] Moutsopoulos HM, Manoussakis MN. Immunopathogenesis of Sjogren's syndrome: "facts and fancy". Autoimmunity. 1989;5(1-2):17-24. doi: 10.3109/08916938909029139. PMID 2519015